CLINICAL TRIAL: NCT04162782
Title: Cross Sectional Study of Iatrogenic Urinary Tract Injuries During Obstetric and Gynecological Operations in Assiut University Women Health Hospital
Brief Title: Urological Injuries During Obstetric and Gynecological Operations
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Kamal Kamel, principal investigator, Assiut University
Other Study IDs: urological injuries
Record Dates: First submitted 2019-11-12; First posted 2019-11-14 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Urologic Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: obstetric and gynaecological surgeries — surgeries for gynecologic and obstetric diseases

SUMMARY:
Iatrogenic urinary tract injuries are more common during obstetric and gynaecological procedures averaging 2.6 per 1000 surgeries . The objective of the study is to estimate the incidence of iatrogenic urinary tract injuries and risk factors during obstetric and gynaecological operations.

Embryologically, the urinary system and genital system have a common origin, so anatomically they are so close that predisposes to iatrogenic trauma to it during obstetric and gynaecological operations. The bladder and distal ureters are the most commonly involved organs. The bladder is a retroperitoneal structure, its trigone rests over the anterior vaginal fornix and the base rests on lower uterine segment and cervix.

DETAILED DESCRIPTION:
Risk factors may contribute to intra-operative bladder injury - include :

1. Prolonged labour with distended bladder.
2. Obstructed labour.
3. Previous cesarean section.
4. previous myomectomy.
5. previous laparotomy.
6. Cases with possibility of altered anatomy, fibrosis or direct extension of disease process as in cases of chronic pelvic inflammatory disease, endometriosis, and large fibroids especially in the broad ligament, previous pelvic surgery, malignancy, previous irradiation and congenital abnormalities of urogenital system.
7. Past history of uterine perforation, septic abortion.
8. In presence of labour, station of the presenting fetal part deeper than or equal to +1, and a large baby were independent risks for a bladder injury during caesarean section.
9. Well effacement and dilatation of cervix (uterine incision may fall over vagina and dissection of bladder from vagina is difficult in compare to lower uterine segment).
10. Preterm cesarean section where lower segment is not well formed.
11. During cesarean hysterectomy.
12. Rupture uterus may also be combined with bladder injuries.
13. Placenta percreta may penetrate the bladder and cause injury.

Urinary tract injury can be diagnosed intraoperative :

1. presence of urine in the operative field.
2. Hematuria
3. Methylene Blue test

ELIGIBILITY:
Inclusion Criteria:

* Women that undergo obstetric or gynecological surgery complicated by urinary tract injury
* Aged 15 years or older
* Elective surgeries
* Good performance status

Exclusion Criteria:

* Not meeting all of the inclusion criteria

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women undergo obstetric or gynecological surgery complicated by urinary tract injury .
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
frequency of iatrogenic urinary tract injuries during obstetric and gynaecological operations. | one month
  frequency of iatrogenic urinary tract injuries during obstetric and gynaecological operations.

REFERENCES:
- [Background] Tarney CM. Bladder Injury During Cesarean Delivery. Curr Womens Health Rev. 2013 May;9(2):70-76. doi: 10.2174/157340480902140102151729. PMID 24876830